CLINICAL TRIAL: NCT04006067
Title: The Impact of Changing Gloves During Cesarean Section on Post-operative Wound Complication. A Single Blind Randomized Controlled Trial
Brief Title: The Impact of Changing Gloves During Cesarean Section on Post-operative Wound Complication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: khalid abd aziz mohamed (Other)
Collaborators: Armed Forces Hospitals, Southern Region, Saudi Arabia (Other Government)
Responsible Party: Sponsor-Investigator, khalid abd aziz mohamed, assistant professor, Benha University
Organization: Benha University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: khalid-shafik
Record Dates: First submitted 2019-06-29; First posted 2019-07-02 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Decreasing Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: changing surgical gloves
- Group B (No Intervention)

INTERVENTIONS:
Other: changing surgical gloves — All the surgical team including surgeons, surgical assists and scrub technicians replaced their outer surgical gloves with a new pair of sterile gloves just prior to abdominal closure.
  Arms: Group A

SUMMARY:
The investigators aim to compare the effect of changing their outer surgical gloves with a new pair of sterile gloves just prior to abdominal closure versus no intervention in the incidence of postoperative wound infections in pregnant women undergoing Caesarean section. The primary outcome is the incidence of any post cesarean wound related complication, including wound seroma, skin separation of at least 1cm, wound infection, or other incisional abnormality requiring treatment within 8 weeks of surgery, while the secondary outcomes are Postoperative fever: defined as greater than 38 degrees Celsius or post cesarean endometritis: defined as a clinical diagnosis, usually involving fever, uterine fundal tenderness, or purulent lochia requiring antibiotic therapy or Combined wound complications and endometritis.

DETAILED DESCRIPTION:
The investigators conduct a prospective randomized study at Department of Obstetrics and Gynecology, AFHSR since April 2019 till October 2019, after approval of the study protocol by the Local Ethical Committee.

Patients undergoing Both elective and emergency cesarean sections and Patients received standard antibiotic prophylaxis within two hours from the procedure or during the procedure in emergency case. All patients received appropriate pre-operative antibiotics, chlorohexidine skin prep except where allergies prohibited, and hair clipping as indicated.

The patients (600) are divided into two groups, Group A (300) during CS the surgical team change their outer surgical gloves with a new pair of sterile gloves just prior to abdominal closure, while in Group B (300) no intervention

ELIGIBILITY:
Inclusion Criteria:

1. Both elective and emergency cesarean sections.
2. Patient received standard antibiotic prophylaxis within two hours from the procedure or during the procedure in emergency case.

Exclusion Criteria:

1. Women with active infection during the procedure.
2. Women did not receive the standard preoperative antibiotic prophylaxis.
3. Women with diagnosis of chorioamnionitis.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of any post cesarean wound related complication | 8 weeks
  including wound hematoma, seroma, skin separation of at least 1cm, wound infection, or other incisional abnormality requiring treatment

CONTACTS AND LOCATIONS:
Locations (1):
- AFHSR, Khamis Mushait, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
will be shared later on